CLINICAL TRIAL: NCT06229301
Title: Artificial Intelligence Assisted Small Incision Lenticule Extraction (SMILE) for Surgical Design and Nomogram Predicting and Related Influencing Factors to Surgical Outcomes
Brief Title: A Study of Artificial Intelligence Assisted Small Incision Lenticule Extraction (SMILE) for Surgical Design and Influencing Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Collaborators: Beihang University (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2023076
Record Dates: First submitted 2023-12-16; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Myopia; Myopic Astigmatism
Keywords: Small-incision Lenticule Extraction; Artificial Intelligence; Nomogram; Refractive Surgery; Myopia Correction
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Experienced-nomogram Group: Patients who underwent Small incision lenticule extraction (SMILE) from March 2014 to October 2018 in Refractive Surgery Center of Tianjin Eye Hospital and had at least three months of postoperative follow-up were included in this group. The Nomogram were based on experience of the surgeon.
- AI-nomogram Group 1: Patients who underwent Small incision lenticule extraction (SMILE) from November 2018 to May 2021 in Refractive Surgery Center of Tianjin Eye Hospital and had at least three months of postoperative follow-up were included in this group. AI-predicted nomogram was obtained and used on patients who underwent surgery.
  Interventions: Procedure: AI-predicted Nomogram
- AI-nomogram Group 2: Patients who underwent Small incision lenticule extraction (SMILE) from January 2023 in Refractive Surgery Center of Tianjin Eye Hospital and had at least three months of postoperative follow-up were included in this group. The datasets used to train AI(Artificial Intelligence) models have been continuously updated for better accuracy since 2018, the newest AI-predicted nomogram was obtained and used on patients who underwent surgery.
  Interventions: Procedure: AI-predicted Nomogram
- Good Surgical Effect and Changes of Biological Parameters: -0.50D < spherical equivalent (SE) < 0.50D
- Poor Surgical Effect and Changes of Biological Parameters: spherical equivalent (SE) <-0.50D or >0.50D

INTERVENTIONS:
Procedure: AI-predicted Nomogram
  Groups: AI-nomogram Group 1; AI-nomogram Group 2

SUMMARY:
The goal of this observational study is to learn about the difference of refractive outcomes between Artificial Intelligence and experienced surgeon predicting Nomogram assist SMILE surgical design and the influenced factors of refractive outcomes in patients who underwent Small Incision Lenticule Extraction(SMILE) at the Refractive Surgery Center of Tianjin Eye Hospital. The main questions it aims to answer are:

* Compare the difference of refractive outcomes between Artificial Intelligence and experienced surgeon predicting Nomogram assist SMILE surgical design
* Analysis the influenced factors of refractive outcomes

DETAILED DESCRIPTION:
In this ambispective observation study, to compare the difference of refractive outcomes between Artificial Intelligence and experienced surgeon predicting Nomogram assist SMILE surgical design and Analysis the influenced factors of refractive outcomes, patients have been continuously recruited and the data can then be used for further case-control and cohort studies.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and older
* Stable refraction over the past 2 years
* Corrected distance visual acuity (CDVA) of 20/25 or better
* Soft contact lens discontinued 2 weeks or longer
* Rigid contact lens discontinued 4 weeks or longer

Exclusion Criteria:

* Abnormal corneal topographic features
* Severe dry eye
* Active keratitis
* Corneal scars
* Keratoconus or suspected keratoconus,
* Glaucoma
* Retina diseases
* History of intraocular or corneal surgery
* Pregnant or lactating women, required chronic systemic corticosteroids or immunocompromised subjects were also excluded from this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This ambispective study included 3246 eyes of 1643 patients with myopia or myopic astigmatism until September 2023. All of patients were accepted the SMILE surgery from May 2014 to June 2023 in Tianjin Eye Hospital. Additional participants will be recruited until September 30, 2024.
  Baseline and postoperative measurements included uncorrected distance visual acuity (UDVA), CDVA, cycloplegic and manifest refraction, slit-lamp and fundus examination, corneal topography and intraocular pressure. Postoperative examinations were scheduled at 1 day, 1 week, 1 month and 3 months. Before surgery, all patients had received 0.5% levofloxacin eyedrops 4 times daily for 3 days.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Diopter | 3 months after small incision lenticule extraction
  Spherical Diopter, cylindrical diopters and axis by Manifest Refraction Test
Uncorrected Distance Visual Acuity (UDVA) | 3 months after small incision lenticule extraction
Corrected Distance Visual Acuity (CDVA) | Before small incision lenticule extraction 3 months after small incision lenticule extraction

SECONDARY OUTCOMES:
Corvis ST Test Result | Before small incision lenticule extraction and 3 months after small incision lenticule extraction
  Using OCULUS Corvis ST Test to obtain biomechanical parameters describing the biomechanical properties of the cornea
Aberration | 3 months after small incision lenticule extraction
  Aberration measured by itrace
Corneal Tomogram | Before small incision lenticule extraction and 3 months after small incision lenticule extraction
  Acquisition of corneal tomograms with the OCULUS Pentacam

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Study Chair — Tiajin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China